CLINICAL TRIAL: NCT00889213
Title: A Prospective Randomized Comparison of Pancreatic Stump Closure Techniques Utilizing an Autologous Falciform Patch and Fibrin Glue Compared to Standard Closure Following Distal Pancreatectomy With or Without Splenectomy
Brief Title: An Evaluation of a New Technique Utilizing a Biologic Glue and Tissue Patch to Seal the Cut Edge of the Pancreas Following Removal of the Tail of the Pancreas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 08D.229
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Pancreatic Fistula; Distal Pancreatectomy Complications; Falciform Patch Pancreatic Closure; Fibrin Glue Pancreatic Closure
Keywords: pancreatectomy; fistula; fibrin glue; falciform patch; surgery; complications
MeSH Terms: conditions — Pancreatic Fistula; Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patch and glue arm (Experimental): Randomized patients to the patch and glue arm will undergo placement of a falciform ligament tissue patch and fibrin glue to the resection margin of the remnant pancreas following distal pancreatectomy
  Interventions: Procedure: Falciform patch and fibrin glue application
- stapled /sutured pancreatic closure (Active Comparator)
  Interventions: Procedure: standard pancreatic closure

INTERVENTIONS:
Procedure: Falciform patch and fibrin glue application — Following standard surgical exploration, the pancreatic gland will be mobilized appropriately to the level of transaction in the pancreatic neck, body or tail. The gland may be divided by stapling device, electrocautery or sharp division. Suture material will be at the discretion of the surgeon but may include absorbable or non-absorbable braided on mono-filament. Those patients randomized to autologous falciform patch will have the falciform membrane harvested. The falciform patch will be laid over the suture line of the resected pancreatic stump and secured to the pancreatic capsule utilizing #4-0 PDS suture placed at 12, 3, 6, and 9 o'clock positions. Fibrin glue (Vitagel) will be utilized to fill the potential space within this membranous capsule. Fibrin glue will be prepared as per standard instructions. Drains will be placed in the splenic bed and/or adjacent to the stump of the pancreas for postoperative fluid evacuation.
  Arms: Patch and glue arm
Procedure: standard pancreatic closure — Following standard surgical exploration, the pancreatic gland will be mobilized appropriately to the level of transaction in the pancreatic neck, body or tail. The gland may be divided by stapling device, electrocautery or sharp division. Suture material will be at the discretion of the surgeon but may include absorbable or non-absorbable braided on mono-filament.
  Arms: stapled /sutured pancreatic closure

SUMMARY:
The purpose of this trial is to determine whether the use of an autologous falciform ligament patch combined with fibrin glue will reduce the rate of pancreatic fistula in patients completing distal pancreatectomy. The hypothesis for the current trial is: Autologous falciform patch closure with fibrin glue will result in a 50% decrease in fistula formation postoperatively. The primary end point will be the development of pancreatic fistula using the ISGPF definition of pancreatic fistula1. (Drain output of any measurable volume of fluid on or after postop day #3 with an amylase content greater than three times serum amylase). Secondary end points will include length of postoperative hospital stay, percutaneous intervention rates, re-operation rates, morbidity to include delayed gastric emptying, wound infection, intraabdominal abscess, postoperative hemorrhage and 30-day mortality.(Bassi C, Dervenis C, Butturini G, et al. Postoperative pancreatic fistula: An international study group (ISGPF) definition. The Journal of Surgery, 2005;138:8-13).

ELIGIBILITY:
Inclusion Criteria:

1. completion of a successful distal pancreatectomy with/without splenectomy
2. patient must have a pancreatic remnant in place
3. there must be a viable falciform ligament for creation of the autologous patch

Exclusion Criteria:

1. patients undergoing total pancreatectomy
2. patients undergoing distal pancreatectomy who have previously completed a right sided resection of the pancreatic head, uncinate and neck
3. failure to sign informed consent
4. pregnant patients
5. patients in whom previous surgery has eliminated the falciform ligament, i.e. previous liver resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2008-08; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Pancreatic fistula development post distal pancreatectomy | 30 days post surgery

SECONDARY OUTCOMES:
Morbidity- wound infection,delayed gastric emptying,abscess formation | 30 day
Mortality | 30 day
Surgical re-intervention/percutaneous interventions | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ernest L Rosato, M.D., Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Carter TI, Fong ZV, Hyslop T, Lavu H, Tan WP, Hardacre J, Sauter PK, Kennedy EP, Yeo CJ, Rosato EL. A dual-institution randomized controlled trial of remnant closure after distal pancreatectomy: does the addition of a falciform patch and fibrin glue improve outcomes? J Gastrointest Surg. 2013 Jan;17(1):102-9. doi: 10.1007/s11605-012-1963-x. Epub 2012 Jul 14. PMID 22798186